CLINICAL TRIAL: NCT06372730
Title: Residual Pulmonary Vascular Obstruction (RPVO) Index Computed with Ventilation/perfusion SPECT/CT Imaging to Predict the Risk of Venous Thromboembolism (VTE) Recurrence in Patients with Pulmonary Embolism (PE)
Brief Title: Residual Pulmonary Vascular Obstruction Index Computed with Ventilation/perfusion SPECT/CT Imaging to Predict the Risk of Venous Thromboembolism Recurrence in Patients with Pulmonary Embolism (PRONOSPECT)
Acronym: PRONOSPECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 29BRC23.0161; 2023-A01566-39 (Other: IDRCB)
Record Dates: First submitted 2024-03-11; First posted 2024-04-18 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Embolism; Venous Thromboembolism
Keywords: venous thromboembolism recurrence
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism | interventions — Ventilation

STUDY DESIGN:
Intervention Model Description: Cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with PE who have been treated with anticoagulant therapy for 3 to 6 uninterrupted months (Experimental): Patients who experienced an objectively proven PE who have been treated initially with anticoagulant therapy for 3 to 6 uninterrupted months (180 - 210 days) and for whom anticoagulation will not be prolonged.
  Interventions: Other: Ventilation/Perfusion Single Photon Emission Computed Tomography (V/Q SPECT/CT)

INTERVENTIONS:
Other: Ventilation/Perfusion Single Photon Emission Computed Tomography (V/Q SPECT/CT) — All patients will undergo a V/Q SPECT/CT scan at inclusion.

SUMMARY:
Major risk after pulmonary embolism (PE) is recurrence, fatal in 10% of patients. Patients with PE can be stratified in 3 groups according to the risk of recurrence : very low risk, high risk or Intermediate risk. Little is known about this last group.

Anticoagulation is efficient to prevent recurrence but is currently not recommended for patient with an intermediate risk of recurrence.

Identifying risk factors of recurrent PE remains a major issue to identify sub-groups of patients who would require lifelong anticoagulation.

In 30-40% of cases, PE patients develop residual pulmonary vascular obstruction (RPVO), which has been found to be associated with an increased recurrence risk. This last observation was mostly reported in patients with unprovoked PE (patients with high risk of recurrence) and RPVO was measured using conventional planar lung scan.

In patients with an intermediate risk of recurrence, the impact of RPVO has been much less studied. In addition, the definition of RPVO was variable according to studies and correlation between RPVO burden and recurrence risk has not been clearly demonstrated. This might be explained by the inherent limitation of RPVO quantification using conventional planar imaging, which is only based on a visual estimation on 2-dimensional images.

Ventilation/Perfusion Single Photon Emission Computed Tomography (V/Q SPECT/CT) is a new method of scintigraphic image acquisition that offers the advantage of 3-dimensional imaging, enabling more accurate and reproducible quantification of RPVO.

The main hypothesis of this study is that in patients with PE at intermediate risk of recurrence, RPVO computed with V/Q SPECT/CT imaging may be an important predictor of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years,
* who experienced an objectively proven PE,
* who have been treated initially with anticoagulant therapy for 3 to 6 uninterrupted months (180 - 210 days) and for whom anticoagulation will not be prolonged.

Exclusion Criteria:

* Unwilling or unable to give written informed consent (protected adults, under tutorship or curatorship)
* Patients deprived of their liberty by a judicial or administrative decision, patients undergoing psychiatric care by virtue of Articles L. 3212-1 and L. 3213-1 who are not covered by the provisions of Article L. 1121-8 and patients admitted to a health or social establishment for purposes other than research
* No Social security affiliation
* Isolated DVT
* Pregnant women,parturients women
* Other indication for anticoagulant therapy (e.g. atrial fibrillation, mechanic valve)
* Life expectancy < 6 months
* Any patients for whom there is a strong indication to treat longer than 6 months: PE provoked by a major persistent factor (e.g. cancer) or Recurrent unprovoked PE
* PE provoked by a major transient risk factor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 665 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Symptomatic recurrent venous thromboembolism (VTE), including objectively confirmed nonfatal symptomatic PE or proximal deep vein thrombosis or fatal PE during a 24-month follow-up after inclusion in the study | From baseline to Month 24
  In case of a suspected VTE or death during follow-up, the study personnel will collect related clinical data on the electronic case report form, and prepare an adjudication file, including symptoms, clinical notes, hospital discharge summary, and results of all diagnostic tests. All suspicion of VTE recurrence will be adjudicated blindly by an independent central Clinical Events Committee.
  To assess the primary objective, RPVO will be defined by a perfusion mismatched defect of at least 5% of the whole lung, corresponding to a segmental defect. SPECT imaging should not be used at inclusion and should not result in proposing prolonged anticoagulation. SPECT images will be numerically stored and interpretation will be later performed independently by two nuclear medicine physicians who will be blinded to clinical history and the patient's outcome. Any difference in interpretation will be resolved by consensus.

SECONDARY OUTCOMES:
Adjudicated symptomatic objectively confirmed recurrent VTE during the follow-up period. | From baseline to Month 24
Percentage of patients with RPVO (as defined by a perfusion defect > 5%) on V/Q SPECT/CT imaging at inclusion in the study. | Inclusion
Different cut-offs of pulmonary vascular obstruction index will be evaluated to predict the risk of VTE recurrence at 2 years, by generating ROC curves | Inclusion
Other predictors of adjudicated symptomatic objectively confirmed recurrent VTE at 2 years including: age | Inclusion
The following score will be computed : HERDOO2 (Hyperpigmentation, Edema, Redness, D-Dimer, Obesity, Old) | Inclusion
  Prediction score of recurrence in patients with unprovoked deep vein thrombosis or pulmonary embolism recurrence in patients with unprovoked PE, (test in patients at intermediate risk of recurrence in this trial). Patient with score of 0 to 1 have a low risk of recurrent VTE, whereas patient with a score of at least 2, have a high risk of recurrence
Potential predictors of RPVO including : demographics | Inclusion
Symptomatic recurrent VTE during a 3 Months follow-up period in patients with suspicion of PE recurrence who has been left untreated based on a negative V/Q SPECT/CT scan | 3 Months follow-up period after the suspicion of PE recurrence
  Symptomatic recurrent VTE including objectively confirmed nonfatal symptomatic PE or proximal DVT or fatal VTE
Dyspnea index will be assessed using mMRC scale (Modified Medical Research Council) | Inclusion and Month 6
  The mMRC scale is a self-assessment tool used to measure the level of impairment caused by breathlessness during daily activities, rated on a scale from 0 to 4.[2] 0, no breathlessness except on strenuous exercise and 4, too breathless to leave the house, or breathless when dressing or undressing.
Quality of life (QoL) will be assessed using PEmb-Qol (Pulmonary Embolism Quality of Life) | Inclusion and Month 6
  The PEmb-QoL is a validated 40-item questionnaire to quantify health-related quality of life in patients having experienced pulmonary embolism (PE). It covers six health dimensions: frequency of complaints, activities of daily living limitations, work-related problems, social limitations, intensity of complaints, and emotional complaints.The PEmb-QoL dimension scores are calculated by taking the mean of the constituting items. Dimension scores are then transformed to a scale from 0-100 to make them comparable across dimensions, with higher scores indicating worse outcome.
Number of Participants with chronic thromboembolic pulmonary hypertension (CTEPH). | From baseline to Month 24
  CTEPH will be defined by a mean pulmonary artery pressure >20 mmHg.
Mortality of all causes. | From baseline to Month 24
Percentage of patients with RPVO (> 5%) on V/Q SPECT/CT imaging using Technegas and Krypton. | Inclusion
The following score will be computed : PADIS-PE score. | Inclusion
  PADIS-PE (score derived from the PADIS study : Prolonged Anticoagulation During eighteen months versus placebo after Initial Six-month treatment for a first episode of idiopathic Pulmonary Embolism randomized trial).
  A higher score indicates a higher risk of recidive.
Other predictors of adjudicated symptomatic objectively confirmed recurrent VTE at 2 years including: gender | Inclusion
Other predictors of adjudicated symptomatic objectively confirmed recurrent VTE at 2 years including: obesity | Inclusion
  Body Mass Index > 30 kg/m2
Other predictors of adjudicated symptomatic objectively confirmed recurrent VTE at 2 years including: D-Dimer | Inclusion
  Measurement of the concentration of plasma D-dimer
Other predictors of adjudicated symptomatic objectively confirmed recurrent VTE at 2 years including: inherited or acquired thrombophilia | Inclusion
  Number of Participants with inherited or acquired thrombophilia
Other predictors of adjudicated symptomatic objectively confirmed recurrent VTE at 2 years including: residual vein thrombosis | Inclusion
  Number of Participants with residual vein thrombosis

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHU Amiens, Amiens, France
  - CHU Angers, Angers, France
  - CHU Brest, Brest, France
  - Hôpital Louis MourierAP-HP, Colombes, France
  - CHD Vendée - La Roche sur Yon, La Roche-sur-Yon, France
  - Kremlin-Bicêtre AP-HP, Le Kremlin-Bicêtre, France
  - CH Les Sables d'Olonne, Les Sables-d'Olonne, France
  - Hegp Ap-Hp, Paris, France
  - CH Quimper, Quimper, France
  - CHU St-Etienne, Saint-Etienne, France
  - CHIC Toulon, Toulon, France
  - HIA Toulon, Toulon, France
  - CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion.
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.